CLINICAL TRIAL: NCT04152317
Title: Comparison Between 200 μg and 800 μg of Misoprostol for Cervical Ripening Prior to Operative Hysteroscopy: Randomized and Quadruple Blind Clinical Trial.
Brief Title: Dose Comparison of Misoprostol for Cervix Ripening Before Operative Hysteroscopy.
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Professor Fernando Figueira Integral Medicine Institute (Other)
Responsible Party: Principal Investigator, Maria da Conceição Farias Souto Maior, Master's Degree, Professor Fernando Figueira Integral Medicine Institute
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Supportive Care
Other Study IDs: MISO.
Record Dates: First submitted 2019-11-02; First posted 2019-11-05 (Actual); Last update posted 2020-10-08 (Actual); Status verified 2020-10

CONDITIONS: Cervix; Open
Keywords: Operative Hysteroscopy; Misoprostol
MeSH Terms: conditions — Uterine Cervical Incompetence | interventions — Misoprostol; Prostaglandins, Synthetic

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Misoprostol 200mcg (Experimental): In this group, the participants will receive 200mcg of misoprostol, single dose, via the vaginal route.
  Interventions: Drug: Misoprostol 200mcg Tab
- Misoprostol 800mcg (Active Comparator): In this group, the participants will receive 800mcg of misoprostol, single dose, via the vaginal route.
  Interventions: Drug: Misoprostol 800mcg Tab

INTERVENTIONS:
Drug: Misoprostol 200mcg Tab — In the misoprostol 200mcg group there will be one tablet of 200mcg and three identical tablets in shape, size and color without pharmacological properties. These four tablets will be single dose administered via vaginal route for each participant.
  Other Names: synthetic prostaglandin
  Arms: Misoprostol 200mcg
Drug: Misoprostol 800mcg Tab — In the misoprostol 800mcg group there will be four tablets of 200mcg. These four tablets will be single dose administered via vaginal route for each participant.
  Other Names: synthetic prostaglandin
  Arms: Misoprostol 800mcg

SUMMARY:
The medication misoprostol is used to facilitate the entry into the uterus of hysteroscopy surgery equipment and this research aims to compare the results of the use of this drug in two different doses trying to find the optimal one.

To perform this work we will use the misoprostol and will perform a questionnaire that will be asked during hospitalization, before, during and the 12hours after the surgery.

The patients who meet the inclusion criteria after signing the Informed Consent Form will be allocated into two groups getting misoprostol 200mcg or misoprostol 800mcg.

DETAILED DESCRIPTION:
Background: Hysteroscopy represents a minimally invasive procedure that has been increasing its adoption in the treatment of many cervical canal and uterine cavity disorders. However, difficulties related to the introduction of the equipment through the cervix are frequent. Although several studies suggest advantages in the cervical preparation with misoprostol, reducing the resistance of the uterine cervix, systematic reviews are unison to indicate the need for clarification on the ideal dose.

Aim: Compare the intra and postoperative results of patients submitted to cervical dilatation for surgical hysteroscopy with previous use of misoprostol at doses of 200mcg or 800mcg for uterine cervix preparation at Recife school hospitals.

Methods: Randomized, quadruple-blind clinical trial with patients who underwent cervical dilatation prior to surgical hysteroscopy at Recife school hospitals, Pernambuco. Patients included will be allocated randomly into two groups. The first group will use misoprostol in the dosage of 200mcg and the second, will use the dosage of 800mcg. Administration, via the vaginal route, will occur 12 hours before performing the operative hysteroscopy. The following variables will be studied: cervical canal width, cervical length, degree of difficulty, duration and failure of cervical dilation, side effects, surgical complications and patient's satisfaction. For statistical analysis, chi-square tests of association, Fisher's exact and Mann-Whitney tests will be used to compare the groups, with an alpha error of less than 5% being considered significant.

Ethical aspects: This study will comply with Resolution 466/12 of the National Health Council and was submitted to and approved by the Professor Fernando Figueira Integral Medicine Institute Research Ethics Committee, beginning only after this approval. All participants will only be included if they voluntarily agree to participate by signing the Free and Informed Consent Form.

There are no conflicts of interest.

ELIGIBILITY:
Inclusion Criteria:

* Patients with indication for operative hysteroscopic.

Exclusion Criteria:

* Patient with contraindications to the use of prostaglandins such as asthma, glaucoma, renal failure, severe heart disease or drug allergy;
* Situations that impede the vaginal administration of medication such as major genital prolapse and virginity;
* Situations that prevent hysteroscopy as major uterine bleeding, diagnosis or suspected topical pregnancy and genital infection such as vaginosis and cervicitis;
* Situations that may influence cervical canal width such as a history of isthmo-cervical incompetence or major cervical surgery like conization or trachelotomy; presence of any structure like uterine fibroid or endometrial polyp inside the cervical canal or though the cervical os; patients on systemic or vaginal estrogen replacement therapy or who have recently used gonadotropin hormone-releasing hormone analogues.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 80 (Actual)
Dates: Start 2019-11-07 (Actual); Primary Completion 2020-09-11 (Actual); Study Completion 2020-09-12 (Actual)

PRIMARY OUTCOMES:
Cervical canal width. | during the surgery
  Maximum size of dilator that passes through the internal os without resistance.

SECONDARY OUTCOMES:
Time required to dilate the cervix to 9mm. | during the surgery
  Time necessary to achieve cervical permeability up to 9mm by introducting the Hegar dilators through the internal os.
Ease of cervical dilation. | during the surgery
  The feeling of ease or difficulty reported by the surgeon while dilating the cervix.
  Evaluated by LIKERT scale. It varies from one to five, one meaning very difficult and five meaning very easy .
Length of the cervix. | during the surgery
  The distance between the external and the internal os measured in centimeters.
Abandonment of the procedure due to cervical dilation failure. | during the surgery
  Impossibility of perform operative hysteroscopy due to difficulty to achieve complete cervical dilation up to 9mm.
Intraoperative complications. | during the surgery
  Complications related to the difficulty of the dilate de cervical canal like uterine perforation, creation of false path, cervical tears and post-dilation bleeding.
Side effects due to the use of the misoprostol. | 24 hours
  Adverse effects as nausea, vomiting, diarrhea, fever, chills, abdominal pain or any other complaint resulting from the use of the medication.
Pain intensity | 24 hours
  The highest level of pain reported by the patient according the Visual Analog Scale evaluated at 3 moments: at the time of hospitalization, at the preoperative time (between medication administration and anesthesia onset) and at the postoperative time (12 hours after the procedure).
Patient satisfaction degree. | 24 hours
  The satisfaction with the medication, reported by the participant. Evaluated by LIKERT scale. It varies from one to five, one meaning less than satisfied and five meaning very satisfied with the drug.

CONTACTS AND LOCATIONS:
Overall Officials: Aurélio Costa, PhD, Study Director — Instituto Materno Infantil Prof. Fernando Figueira
Locations (1):
- Maria da Conceição Souto Maior, Recife, Pernambuco, Brazil

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Maior MDCFS, Souza ASR, Souza GFA, da Costa AAR. Comparison between 200 mug and 800 mug of vaginal misoprostol for cervical ripening before operative hysteroscopy: A randomized controlled trial. Int J Gynaecol Obstet. 2022 Jul;158(1):205-212. doi: 10.1002/ijgo.13984. Epub 2021 Nov 3. PMID 34695232